CLINICAL TRIAL: NCT04576065
Title: Randomized Controlled Trial of the Wake Forest Post-ICU Telehealth (WFIT) Program
Brief Title: Wake Forest Post-ICU Telehealth (WFIT) Program
Acronym: WFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00068761
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-05

CONDITIONS: Critical Illness
Keywords: post-ICU; post-intensive care; ICU recovery; critical illness recovery
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: usual care group compared to intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients randomized to usual care will follow-up with primary care providers and specialists as recommended by hospital providers, or seek medical care as needed after hospital discharge.
- Intervention (Experimental): Patients randomized to intervention will have 6 months of access after hospital discharge for telehealth visits with a nurse practitioner and an activity tracker providing data to the nurse practitioner about subject's daily level of activity.
  Interventions: Other: WFIT

INTERVENTIONS:
Other: WFIT — access to nurse practitioner for telehealth visits and activity monitor for 6 months after hospital discharge
  Arms: Intervention

SUMMARY:
Wake Forest Post-Intensive Care Unit Telehealth (WFIT) program consists of a nurse practitioner who has access to daily activity data as well as telehealth capabilities for 6 months post-hospital discharge in order to improve the post-critical illness care of patients. The study team expects that this program will reduce costs to patients. Through this intervention the study team hopes to improve quality of life, patient satisfaction, reduce readmissions and ER visits, and reduce mortality. The study team will perform a formal randomized controlled trial with a cost-effectiveness analysis to demonstrate its value.

DETAILED DESCRIPTION:
Wake Forest Baptist Health (WFBH) discharges over 1,000 patients annually after a critical illness such as septic shock and/or acute respiratory failure. This number is expected to be even higher due to the ongoing coronavirus pandemic. To try to bridge this gap, the Wake Forest Intensive Care Unit (ICU) Recovery Clinic was created in 2014. WFBH ICU Recovery Clinic (1 of ~15 nationwide) uses a multidisciplinary approach to transition care for ICU survivors back to Primary Care Physicians (PCPs). However, currently only about 5% of patients leaving the ICU who had respiratory failure and/or septic shock and may benefit from follow-up. In addition, patients seen in WFBH Recovery Clinic typically are only seen one time and then return to the care of their PCPs.

Poor physical function following critical illness is associated with hospital readmissions and mortality. However, barriers to post-ICU follow-up are common and include financial concerns as well as transportation barriers. Additionally, the Wake Forest ICU Recovery Clinic only sees patients once in the post-critical illness period, despite the fact that post-ICU morbidity remains high for at least six months following discharge. Finally, data demonstrates availability of internet services on a daily basis to the vast majority of the population (79% total of NC Congressional Districts 5, 6, and 13 in 2013; 68% in a random sample of 28 medical ICU patients). Taken together, this prompts the study team to propose this Wake Forest Post-ICU Telehealth (WFIT) program of a nurse practitioner who has access to daily activity data as well as telehealth capabilities in order to improve the post-critical illness care of these patients. The study team expects that this program will reduce costs to patients. Through this intervention the study team hopes to improve quality of life, patient satisfaction, reduce readmissions and ER visits, and reduce mortality. The study team will perform a formal randomized controlled trial with a cost-effectiveness analysis to demonstrate its value.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Wake Forest Baptist Health medical Intensive Care Unit (ICU)
* North Carolina Residents
* ICU Diagnosis: Sepsis and/or acute respiratory failure defined by assisted ventilation (includes mechanical ventilation, Bilevel Positive Airway Pressure (BIPAP), Continuous Positive Airway Pressure (CPAP), or requiring > 15 Liter of supplemental oxygen
* Consent to enrollment in the study
* Survive to hospital discharge

Exclusion Criteria:

* >2 Hospitalizations in the past year.
* Admitted from hospice, a skilled nursing facility or Long-Term Acute Care Hospital (LTACH).
* Discharge to a Skilled Nursing Facility or LTACH or Hospice. We will permit enrollment of patients who are discharged to acute rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Incremental Net Benefit (INB) Cost Effectiveness | 6 months post hospital discharge
  Determine if the WFIT Program is cost-effective by measuring INB in the intervention arm (WFIT program) compared to an attention control arm.
  Incremental net benefit ($) = [Change in Quality of Adjusted Life Year (QALY) *100,000] - [Change in health care spending]
  INB is defined as the difference between change in quality of life evaluated at monetary valuation of 1 QALY (currently $100,000) and change in health care spending. Using this measure, even if WFIT does not affect patient quality of life, then INB will equal the reduction in health care spending.

SECONDARY OUTCOMES:
Number of Emergency Room (ER) Visits | 6 months post hospital discharge
  evaluated monthly through to 6 months.
Number of hospital readmissions | 6 months post hospital discharge
  Readmissions to a hospital evaluated monthly through to 6 months.
Mortality Rate | Through 6 months post hospital discharge
Patient Satisfaction Questionnaire 18 (PSQ-18) | 6 months post hospital discharge
  Satisfaction with care evaluated monthly through to 6 months. Scores range from 18-90 with a higher score denoting more satisfaction.
Euro Quality of Life, 5 Dimension, 5 Level (EQ-5D-5L) Questionnaire | 6 months post hospital discharge
  Quality of life evaluated monthly through to 6 months. Scores range from 5-25 with higher scores indicating poorer health status.

CONTACTS AND LOCATIONS:
Overall Officials: Clark Files, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakhru RN, Flores L, Cain JM, Province V, Fanning J, Rawal H, Bundy R, Obermiller CS, Moses A, Dharod A, Abdelfattah L, Hanchate A, Files DC. A Randomized Controlled Trial of a Post-ICU Telehealth Care Model (WFIT). Am J Respir Crit Care Med. 2025 Sep;211(9):1662-1670. doi: 10.1164/rccm.202411-2167OC. PMID 40532205

DOCUMENTS (1):
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT04576065/ICF_000.pdf